CLINICAL TRIAL: NCT01471834
Title: Neo Non-Randomized Hypertension Study
Brief Title: Verification of the Efficacy and Safety of the BAROSTIM NEO System in the Treatment of Drug Resistant Hypertension
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 360016
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Device and Medical Management (Experimental): Participants will be implanted with the BAROSTIM NEO System and will continue to receive optimal, stable, Guideline Directed Medical Therapy (GDMT) for heart failure (American Heart Association [AHA] / American College of Cardiology [ACC] guidelines), including drugs to be determined by the subject's physician. Drug types include: Loop Diuretics, Thiazide Diuretics, Potassium-sparing Diuretics, Sequential Nephron Blockade, ACE Inhibitors, ARBs, ARNI, Aldosterone Antagonists, Beta Blockers and Hydralazine and Isosorbide Dinitrate.
  Interventions: Device: BAROSTIM NEO System; Drug: Medical Management

INTERVENTIONS:
Device: BAROSTIM NEO System
  Other Names: XR-1 System; Neo System
Drug: Medical Management

SUMMARY:
To assess the long-term safety and efficacy of the BAROSTIM NEO System in trial (NCT01471834) participants.

DETAILED DESCRIPTION:
The Neo Non-Randomized Hypertension Study is a non-randomized, open-label, verification study in participants diagnosed with drug resistant hypertension, defined as medical treatment failure for hypertension defined as office cuff systolic blood pressure (SBP) ≥ 140 mmHg despite being prescribed to at least three antihypertensive medications, including a diuretic, in accordance with the AHA guidelines.

Participants should remain on their prescribed anti-hypertensive medications and same dosing schedule for the duration of the study unless investigators determine medically necessary changes are needed. Additionally, every effort should be made to maintain adequate rate control for subjects with atrial fibrillation throughout the duration of the study.

All (Canadian) participants are now in long term follow-up and are required to have at least one annual visit.

Parameters assessed during long-term follow-up visits:

* Physical Assessment
* Office Cuff Blood Pressure
* Subject Medications
* Serious adverse events

ELIGIBILITY:
Inclusion Criteria:

* Actively participating in the Neo Non-Randomized Hypertension Study.
* Have signed a revised approved informed consent form for continued participation in this study.

Exclusion Criteria:

* Treating physician decision that the subject should not continue with therapy.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To access long-term adverse events in participants implanted with the BAROSTIM NEO System. | For the duration of the study, up to 10 years.
  Ascertain the type, frequency, severity and timing of long-term adverse events in participants implanted with the device, while providing a viable treatment option to participants currently implanted with CVRx's BAROSTIM NEO System.

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Haller, MD, Principal Investigator — Hannover Medical School
Locations (9):
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - University of Alberta - Edmonton, Edmonton, Alberta
  - London-Lawson Health Research Institute, London, Ontario
- Germany (5):
  - University Hospital Cologne, Cologn
  - University Hospital Duesseldorf, Düsseldorf
  - Goettingen-Georg August University, Göttingen
  - Midizinische Hochschule Hannover, Hanover
  - Klinkum St. George Leipzig, Leipzig
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Wachter R, Halbach M, Bakris GL, Bisognano JD, Haller H, Beige J, Kroon AA, Nadim MK, Lovett EG, Schafer JE, de Leeuw PW. An exploratory propensity score matched comparison of second-generation and first-generation baroreflex activation therapy systems. J Am Soc Hypertens. 2017 Feb;11(2):81-91. doi: 10.1016/j.jash.2016.12.003. Epub 2016 Dec 16. PMID 28065708